CLINICAL TRIAL: NCT01816048
Title: A Pharmacodynamic Study Using NaF PET/CT Imaging to Assess Treatment Responsiveness to TAK-700 in Patients With Metastatic Castrate Resistant Prostate Cancer to Bone
Brief Title: NaF Positron Emission Tomography/Computed Tomography (PET/CT)Imaging to Assess Treatment Responsiveness to TAK-700 in Patients With Castrate Resistant Prostate Cancer (CRPC) With Bone Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study supporter (Takeda) ended study drug for prostate cancer; enrollment ended prematurely.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO12810; 2012-1107 (Other: Institutional Review Board); NCI-2013-01081 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-12

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: prostate, prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAK-700 (Experimental): TAK-700 will be administered at 300 mg orally (PO)twice daily (BID) continuously on 28-day treatment cycles.
  The most common way of assessing bone metastasis is planar bone scintigraphy or single photon emission computed tomography (SPECT), though both lack high spatial resolution and thus make small metastases detection inaccurate. Positron emission tomography (PET) is a successful imaging modality with a higher resolution than SPECT, but has not been widely adopted in bone imaging. One of the most promising PET imaging agents for detection of bone metastasis is 18F-Sodium Fluoride (Fluorine F 18 Sodium Fluoride, or NaF). NaF uptake is characterized by high and rapid bone uptake accompanied by very rapid blood clearance, which results in a high bone-to-background ration in a short time.
  Interventions: Drug: TAK-700; Radiation: Fluorine F 18 Sodium Fluoride; Procedure: Positron Emission Tomography; Procedure: Computed Tomography

INTERVENTIONS:
Drug: TAK-700 — TAK-700 will be administered at 300mg twice per day on 28-day continuous cycles
  Other Names: orteronel
Radiation: Fluorine F 18 Sodium Fluoride — Undergo NaF F18 PET/CT scan
  Other Names: 18 F-NaF; F-18 NaF
Procedure: Positron Emission Tomography — Undergo 18F NaF PET/CT scan
  Other Names: PET
Procedure: Computed Tomography — Undergo 18F NaF PET/CT scan
  Other Names: CT; CAT Scan

SUMMARY:
The purpose of this study is to assess whether NaF PET/CT scans can be used to evaluate treatment response in bone metastases in subjects with prostate cancer treated with the investigational drug, TAK-700.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18 years or older
* Voluntary written consent
* Histologically proven adenocarcinoma of the prostate
* Evidence of radiographic bone metastases
* May have received prior chemotherapy for metastatic disease, but prior chemotherapy is not a requirement for eligibility
* Eastern Cooperative Oncology Group performance status 0-2
* Serum testosterone level is less than or equal to 50 ng/dL
* Has undergone orchiectomy or plan to continue receiving gonadotropin releasing hormone (GnRH) analogue therapy
* Adequate organ function as measured by screening laboratory values specified in the protocol
* Must agree to use appropriate contraceptives prior to study procedures, during duration of study participation and for 4 months after last dose of TAK 700
* Must be able to lie flat for greater than or equal to 30 minutes during PET/CT imaging
* Screening calculated ejection fraction of greater than or equal to 50% by multigated radionuclide angiography (MUGA) scan or Echocardiogram

Exclusion Criteria:

* Received Strontium-89, Samarium-153, or other radioisotope within 3 months of registration
* history of allergic reactions attributed to compounds similar to sodium fluoride F-18 (NaF)
* history of seizure disorder
* Known history of brain metastases
* Concurrent treatment with any herbal products within 7 days of study entry
* Received radiotherapy less than or equal to 4 weeks prior to registration
* Known hypersensitivity to TAK-700 or related compounds
* Prior therapy for treatment of metastatic castrate resistant prostate cancer with any androgen biosynthesis inhibitor or androgen signaling pathway inhibitor such as: enzalutamide (MDV-3100), abiraterone, ketoconazole, or aminoglutethimide
* Current bladder neck outlet obstruction
* Current spinal cord compression
* Current bilateral hydronephrosis
* History of adrenal insufficiency
* History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias (over grade 2), thromboembolic events, or any other cardiac condition within 6 months prior to first dose of study drug.
* Uncontrolled high blood pressure
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Major surgery less than or equal to 4 weeks before the first dose of study drug
* Serious infection less than or equal to 2 weeks before the first dose of study drug
* Known gastrointestinal (GI) disease or GI procedure that could interfere with oral absorption or tolerance of TAK-700, including difficulty swallowing capsules

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justine Y Bruce, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- TAK-700: TAK-700 was administered at 300 mg orally (PO)twice daily (BID) continuously on 28-day treatment cycles.
  TAK-700: TAK-700 will be administered at 300mg twice per day on 28-day continuous cycles
  Fluorine F 18 Sodium Fluoride: Undergo NaF F18 PET/CT scan
  Positron Emission Tomography: Undergo 18F NaF PET/CT scan
  Computed Tomography: Undergo 18F NaF PET/CT scan
Period: Overall Study
Arm/Group | TAK-700
Started | 8
Completed | 2
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | TAK-700
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Maximum NaF PET/CT Standardized Uptake Values
Description: To measure changes in NaF PET/CT standardized uptake values (SUVmax) from prior to dosing with Tak-700 to12 weeks after starting treatment with TAK-700. Value at three months minus value at baseline.
Time Frame: Baseline and 3 months
Population: The study closed early so only 8 of 20 planned were enrolled and of the 8, only 4 completed the week 12 scan.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 4
Participants
  SUVmax decrease | 3
  SUVmax increase | 1

2. Primary Outcome: Number of Participants With Change in Prostate Specific Antigen (PSA) Response Rate
Description: Measure prostate specific antigen (PSA) response rate in patients treated with TAK700, as measured by a decline in the PSA level from baseline to the month 3 assessment according to the Prostate Cancer Clinical Trials Working Group (PCWG2), at least a 50% decrease from baseline. Percent increase or decrease from month three compared to baseline.
Time Frame: Baseline and 3 months
Population: Study closed early and only 8 of planned 20 enrolled. Four subjects came off study prior to the three month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 4
Participants
  PSA decline >= 50% | 3
  PSA decline =< 50% | 1

3. Secondary Outcome: Number of Subjects Who Experience Adverse Events While on Treatment With TAK 700
Description: The number of subjects experiencing adverse events per CTCAE 4.0 while on treatment.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Groups:
- TAK-700: TAK-700 will be administered at 300 mg orally (PO)twice daily (BID) continuously on 28-day treatment cycles.
  TAK-700: TAK-700 will be administered at 300mg twice per day on 28-day continuous cycles
  Fluorine F 18 Sodium Fluoride: Undergo NaF F18 PET/CT scan at screen, week 4-8 and week 12
Arm/Group | TAK-700
Number analyzed (Participants) | 8
participants | 8

4. Secondary Outcome: Number of Patients With a Measurable Change in PSA Kinetics With TAK700 From Baseline to Off Treatment
Description: Stable: no change in PSA kinetics Decrease: less than baseline Increase: greater than baseline
  PSA data was gathered at baseline and off treatment.
Time Frame: Up to 14 months
Population: Due to study closing early only 8 of planned 20 patients enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 8
Participants
  Stable | 1
  Decrease in PSA | 3
  Increase in PSA | 4

5. Secondary Outcome: Number of Participants With Changes in NaF PET/CT Results in Response to TAK700
Description: This is an exploratory endpoint as we are planning to identify other new parameters during the PET/CT scanning that may be more predictive of response (such as SUV volume, or dynamic changes during the scanning period). Changes in results at week 12 compared to baseline. Value at 12 weeks minus value at baseline.
Time Frame: At baseline and 12 weeks
Population: Due to study closing early only 8 of planned 20 patients enrolled and only 4 of the 8 subjects enrolled completed the week 12 scan.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 4
Participants
  Increase in SUV total | 1
  No change | 1
  Decrease in SUV total | 2

6. Secondary Outcome: Compare Changes on NaF PET/CT After Treatment With TAK700 With Standard Clinical Outcomes Including PSA Doubling Time, Response Evaluation Criteria in Solid Tumors (RECIST), and Radiographic Progression Free Survival.
Time Frame: Approximately 24 months
Population: Due to study closing early, only 8 of planned 20 patients enrolled. Data for this endpoint was not obtained.
Arm/Group | TAK-700
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With a Change in the Number of Circulating Tumor Cells Using One or More Methods (Epispot)
Description: Baseline compared to 12 weeks. Value at three months minus value at baseline.
Time Frame: At baseline and 12 weeks
Population: Due to study closing early only 8 of 12 patients enrolled, and only 5 subjects obtained a week 12 CTC test.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 5
Participants
  Increase in circulating tumors | 2
  Decrease in circulating tumors | 3

8. Secondary Outcome: Number of Participants With Change in the Number of Circulating Tumor Cells Using the Cell Search System (Veridex, LLC) Obtained Prior to Beginning Treatment With TAK 700, After Completing One Cycle and After Completing 3 Cycles
Description: Change from baseline to one month and three month.
Time Frame: At baseline, one month, three months
Population: Due to study closing early only 8 of planned 20 enrolled. All subjects completed one month of treatment; only 4 subjects completed the week 12 scan.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 8
Participants
  Cycle 1 (one month): Increase in circulating tumors | 2
  Cycle 1 (one month): Decrease in circulating tumors | 5
  Cycle 1 (one month): No change | 1
  Cycle 4 (three months): number analyzed (Participants) | 4
  Cycle 4 (three months): Increase in circulating tumors | 1
  Cycle 4 (three months): Decrease in circulating tumors | 1
  Cycle 4 (three months): No change | 2

9. Secondary Outcome: PSA Response Rate and Circulating Tumor Cell Counts of Subjects Receiving TAK700 to NaF PET/CT Imaging Results
Time Frame: Baseline, one month, 2 months, 3 months
Population: Data was not collected for this outcome measure.
Arm/Group | TAK-700
Number analyzed (Participants) | 0

10. Primary Outcome: Number of Participants With a Change in Total NaF PET/CT Standardized Uptake Values
Description: To measure changes in NaF PET/CT standardized uptake values (SUV total) from prior to dosing with Tak-700 to12 weeks after starting treatment with TAK-700. Percent change from three months to baseline; value at three months minus value at baseline.
Time Frame: Baseline and 3 months
Population: The study closed early so only 8 of 20 planned were enrolled and of the 8, only 4 completed the week 12 scan.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-700
Number analyzed (Participants) | 4
Participants
  SUV total increase | 1
  SUV total decrease | 2
  SUV total no change | 1

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Description: All patients were followed for adverse events for at least 30 days after the last dose of TAK-700, or before the initiation of another systemic antineoplastic therapy, whichever came first. Adverse events were assessed at all study visits and follow ups.
Arm/Group | TAK-700
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-700 (N=8)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Nerve impingement (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
sudden death (General disorders) | 1 (1) — Patient died at home no cause of death determined.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-700 (N=8)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Allergic rhinitis (Immune system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Disuria (Renal and urinary disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (6)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Injury, arm (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (14)
Pain (General disorders) | 3 (8)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal calculi (Renal and urinary disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
neoplasms benigh, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — squamous cell skin right ear
Stomach pain (Gastrointestinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 3 (3)
nerve impingement (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No